CLINICAL TRIAL: NCT01942291
Title: Short-term Effect of Extended-release Niacin With and Without the Addition of Laropiprant on Endothelial Function
Brief Title: Short-term Effect of Extended-release Niacin on Endothelial Function.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, Professor, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Unicamp845/2011
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Hypoalphalipoproteinemia
Keywords: Niacin; Endothelial function; Laropiprant; HDL
MeSH Terms: conditions — Hypoalphalipoproteinemias | interventions — Niacin; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Niacin/Laropiprant (Experimental): Extended-release niacin 1g/day associated with Laropiprant 1g/20mg (ERN/LRPT, Cordaptive, Merck, Sao Paulo, Brazil)
  Interventions: Drug: Niacin
- Niacin (Experimental): Extended-release niacin 1g/day alone (ERN, Metri, Libbs Farmaceutica, Sao Paulo, Brazil)
  Interventions: Drug: Niacin

INTERVENTIONS:
Drug: Niacin — The study was randomized, double-blind, controlled, using a 2-way crossover design with both treatment periods and washout time lasting 7 days. Subjects were allocated by simple randomization to extended-release niacin 1g/day alone (ERN, Metri, Libbs Farmacêutica, São Paulo, Brazil) or niacin associated with LRPT 1g/20mg (ERN/LRPT, Cordaptive, Merck, São Paulo, Brazil).
  Other Names: Nicotinic acid; Vitamin B3

SUMMARY:
Individuals with reduced plasma concentration of high-density lipoprotein (HDL) cholesterol are more susceptible to oxidative stress and often present reduced endothelial function, which has been mainly related to this susceptibility. Studies in animal and cell models have demonstrated that niacin activates both GPR-109A in leukocytes and heme oxygenase-1 (HO-1) pathway promoting strong anti-inflammatory and anti-oxidative effects. . In this context, the aim of this study was to investigate the short-term effect of niacin on endothelial function and verify the existence of interaction of PGD2 receptor antagonist, i.e. laropiprant (LRPT), in subjects with low HDL-cholesterol (HDL -C).

DETAILED DESCRIPTION:
Study design and treatments The study was randomized, double-blind, controlled, using a 2-way crossover design with both treatment periods and washout time lasting 7 days. Subjects were allocated by simple randomization to extended-release niacin 1g/day alone (ERN, Metri, Libbs Farmacêutica, São Paulo, Brazil) or niacin associated with LRPT 1g/20mg (ERN/LRPT, Cordaptive, Merck, São Paulo, Brazil). Medications were kindly supplied by Libbs and Merck. Plasma samples and brachial artery reactivity were obtained at baseline, 7th day of treatment 1, 7th day after washout and 7th day of treatment 2.

Study Measurements The following blood measurements were performed using the Modular Hitachi system and Roche Diagnostics (Mannheim, Germany) reagents: glucose (GOD-PAP), triglycerides (TG)(GPO-PAP), HDL-C (HDL-C plus 3rd generation) and C-reactive protein (CRP) (high-sensitivity CRP, Cardiophase, Dade Behring, Marburg, Germany). LDL cholesterol was calculated by the Friedewald formula. HDL size was measured by laser scattering (Zetasizer - Nanoseries DTS 1060, Malvern Instruments, Worcestershire, UK). Total and direct bilirrubin was measured by the Jendrassik-Grof method (Roche/Hitachi analyzer).

The cholesteryl ester transfer protein activity was measured by an endogenous assay. Aliquots of the whole plasma (in which LCAT activity was inhibited by DTNB 9 μL/mL) were added to HDL-[3H]cholesteryl ester fractions and simultaneously incubated at 4°C and 37°C for 4h. Apo-B containing lipoproteins, present in the incubation mixture, were then precipitated; the CE radioactivity in the supernatant represented the net rate at which CE mass was transferred and values expressed as percent of [3H] cholesteryl ester transferred/4 hours depended upon the plasma concentrations of HDL, TG-rich lipoproteins and CETP simultaneously.

Endothelial-dependent vasodilation was assessed by ischemia-induced reactive hyperemia. Briefly, after 12-hour overnight fasting patients were examined at 8 a.m. in a quiet room at 22ºC by using a ultrasound equipment Vivid i (GE Healthcare, Wauwatosa, WI, USA) with a high-resolution (up to 13 MHz) vascular probe (12l-RS, GE Healthcare, Wauwatosa, WI, USA) in B-mode. The cardiac cycles were monitored simultaneously by electrocardiography coupled to the equipment. Flow-mediated dilation (FMD) was assessed after 5-minutes inflation of a cuff placed below the transducer, 50 mm Hg above the systolic blood pressure. Two-dimensional images of the brachial artery were obtained during 5 minutes from the longitudinal axis approximately 5-10 cm above the antecubital fossa. The maximum expansion of the diameter of the brachial artery was measured in triplicate at the peak of the T wave of the cardiac cycle before the interruption of the flow and post deflation.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic individuals
* plasma HDL-C levels <40 mg/dL

Exclusion Criteria:

* symptomatic atherosclerotic disease
* diabetes
* liver disease
* renal disease
* thyroid dysfunction
* indication for or use of lipid-lowering treatment in the last six months
* use of anti-inflammatory treatment in the last 30 days
* current or previous diagnosis of cancer or immune inflammatory diseases
* chronic obstructive pulmonary disease
* infectious disease manifested in the last 3 months
* body mass index ≥ 26 kg/m2

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The short-term effect of niacin on endothelial function. | 7 days
  Endothelial-dependent vasodilation was assessed by ischemia-induced reactive hyperemia of the brachial artery by using an ultrasound equipment

SECONDARY OUTCOMES:
Plasma C-reactive protein levels | 7 days
  Systemic inflammatory activity as estimated by the plasma concentration of C-reactive protein
HDL-C and HDL size | 7 days
  Plasma concentration of high-density lipoprotein (HDL) cholesterol and HDL size

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, PhD, Principal Investigator — University of Campinas
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Nasser Figueiredo V, Vendrame F, Colontoni BA, Quinaglia T, Roberto Matos-Souza J, Azevedo Moura F, Coelho OR, de Faria EC, Sposito AC. Short-term effects of extended-release niacin with and without the addition of laropiprant on endothelial function in individuals with low HDL-C: a randomized, controlled crossover trial. Clin Ther. 2014 Jun 1;36(6):961-6. doi: 10.1016/j.clinthera.2014.03.012. Epub 2014 Apr 24. PMID 24768191